CLINICAL TRIAL: NCT06893497
Title: Does Low-level Laser Therapy Protocol Affect the Efficacy of Treatment of Inferior Alveolar Nerve Injury After Maxillofacial Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Halenur Ateş, DDS, Karadeniz Technical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/8
Record Dates: First submitted 2025-02-08; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Inferior Alveolar Nerve Injuries
MeSH Terms: conditions — Mandibular Nerve Injuries | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with different sessions, start time and cause of IAN injury were compared. (Experimental): Low level laser therapy was applied to all patients.
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Device: Low Level Laser Therapy — In this study, which had more patients than other studies, different parameters were evaluated to determine the protocol of LLL therapy. These parameters were the cause of IAN injury, number of sessions, time of treatment start and period of follow-up.

SUMMARY:
Dear Patient, Dear Parent / Guardian; This consent form has been prepared to enlighten you about the nature of the diagnosis and treatment methods that have been explained to you/patient and will be applied, the expected benefits of the procedures, possible side effects, alternative diagnosis and treatment options and their characteristics, and the consequences that may arise if these procedures are not performed and to obtain your consent. By reading and signing this form, you declare that you have been informed about the procedure and that you freely consent to the procedure. You can ask your doctor about the points you do not understand in the form. Please bring this form with you on the day of your appointment and hand it to your doctor.

WHAT YOU NEED TO KNOW DIAGNOSIS AND PROCEDURE: Low-level laser therapy will be applied for the treatment of sensory impairment resulting from maxillofacial surgery.

WHO WILL PERFORM YOUR PROCEDURE? This procedure will be performed by the physicians working in Karadeniz Technical University Faculty of Dentistry, Oral, Dental and Maxillofacial Surgery. I also accept that KTU Faculty of Dentistry is an educational institution and that my treatment can be used to contribute to the education of interns and that they can participate in my operation.

EXPECTED BENEFITS OF THE PROCEDURE To contribute to the nerve regeneration of the patient whose quality of life has deteriorated due to sensory damage.

PROBLEMS THAT MAY BE ENCOUNTERED IF THE PROCEDURE IS NOT PERFORMED There is no risk associated with low-level laser treatment.

ALTERNATIVES TO THE PROCEDURE, IF ANY: There is no alternative treatment.

possible risks and complications of the procedure Treatment approaches to nerve injuries are divided into two as surgical and non-surgical treatment approaches. Surgical treatment approaches include decompression, resection of neuroma, internal neurolysis, neurorrhaphy, nerve grafts and intubation techniques. However, since there is a risk of complications after surgical treatment, non-surgical treatment approaches are primarily preferred. Non-surgical treatment approaches include pharmacological treatment, acupuncture, moxibustion and low-level laser (DSL) treatment.

ESTIMATED DURATION OF THE PROCEDURE: 15-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral or bilateral inferior alveolar nerve damage caused by maxillofacial surgery and receiving DESL treatment
2. Patients with a follow-up period of at least 6 months
3. Patients whose diagnosis has been confirmed by clinical neurosensory testing
4. Patients with complete study data and follow-up
5. Patients who have not previously undergone any microsurgical or conservative treatment in the head and neck region due to nerve damage
6. Patients without known neurological disease that may affect the study results
7. Patients without active infection (pain, temperature increase, redness, edema, loss of function, etc.) or pathological findings (tumour, cyst, etc.) in the relevant area were included.

Exclusion Criteria:

1. Patients with nerve damage due to other reasons (pathology, infection, etc.) before maxillofacial surgery
2. Patients with lingual nerve damage
3. Patients with known neurological disease that may affect the study results
4. Patients with missing data or patients who cannot be followed up
5. Pregnant patients were not included in the study.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
the Visual Analog Scale (VAS) | up to 2 years
  All patients underwent preoperative and postoperative clinical neurosensory testing (CNT), comprising three levels of evaluation. Level A: two-point discrimination, where the minimum distinguishable distance (15 mm, 10 mm, and 5 mm) was measured using slight skin pressure. Level B: light touch assessment, where a blunt-tipped tool was applied to 10 points on the lower lip, recording detected stimuli. Level C: pin-prick nociception, where forceps compression assessed pain perception at 10 points. A subjective neurosensory deficit assessment was conducted using the Visual Analog Scale (VAS), a 100 mm horizontal line ranging from 0 (no sensation) to 100 (normal sensation), with descriptors at both ends.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Jan 2019 - Jan 2023

REFERENCES:
- [Result] Guarini D, Gracia B, Ramirez-Lobos V, Noguera-Pantoja A, Sole-Ventura P. Laser Biophotomodulation in Patients with Neurosensory Disturbance of the Inferior Alveolar Nerve After Sagittal Split Ramus Osteotomy: A 2-Year Follow-Up Study. Photomed Laser Surg. 2018 Jan;36(1):3-9. doi: 10.1089/pho.2017.4312. Epub 2017 Oct 12. PMID 29022844
- [Result] Favaro-Pipi E, Feitosa SM, Ribeiro DA, Bossini P, Oliveira P, Parizotto NA, Renno AC. Comparative study of the effects of low-intensity pulsed ultrasound and low-level laser therapy on bone defects in tibias of rats. Lasers Med Sci. 2010 Sep;25(5):727-32. doi: 10.1007/s10103-010-0772-2. Epub 2010 Jun 3. PMID 20521077
- [Result] Miloro M, Repasky M. Low-level laser effect on neurosensory recovery after sagittal ramus osteotomy. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2000 Jan;89(1):12-8. doi: 10.1016/s1079-2104(00)80006-2. PMID 10630935
- [Result] Moore KC., Hira N., Kumar PS., Jayakumar CS., Ohshiro T. A Double Blind Crossover Trial of low Level Laser Therapy in the Treatment of Postherpetic Neuralgia. Laser Ther 2004;14:61-4. Doi: 10.5978/ISLSM.14.0_61.
- [Result] Kahraman SA. Low-level laser therapy in oral and maxillofacial surgery. Oral Maxillofac Surg Clin North Am. 2004 May;16(2):277-88. doi: 10.1016/j.coms.2004.02.002. No abstract available. PMID 18088730
- [Result] Sun G, Tuner J. Low-level laser therapy in dentistry. Dent Clin North Am. 2004 Oct;48(4):1061-76, viii. doi: 10.1016/j.cden.2004.05.004. PMID 15464564
- [Result] Mohajerani SH, Tabeie F, Bemanali M, Tabrizi R. Effect of Low-Level Laser and Light-Emitting Diode on Inferior Alveolar Nerve Recovery After Sagittal Split Osteotomy of the Mandible: A Randomized Clinical Trial Study. J Craniofac Surg. 2017 Jun;28(4):e408-e411. doi: 10.1097/SCS.0000000000002929. PMID 28538060
- [Result] Ozen T, Orhan K, Gorur I, Ozturk A. Efficacy of low level laser therapy on neurosensory recovery after injury to the inferior alveolar nerve. Head Face Med. 2006 Feb 15;2:3. doi: 10.1186/1746-160X-2-3. PMID 16480503
- [Result] Robinson PP, Loescher AR, Yates JM, Smith KG. Current management of damage to the inferior alveolar and lingual nerves as a result of removal of third molars. Br J Oral Maxillofac Surg. 2004 Aug;42(4):285-92. doi: 10.1016/j.bjoms.2004.02.024. PMID 15225944
- [Result] Esteves Pinto Faria P, Temprano A, Piva F, Sant'ana E, Pimenta D. Low-level laser therapy for neurosensory recovery after sagittal ramus osteotomy. Minerva Stomatol. 2020 Jun;69(3):141-147. doi: 10.23736/S0026-4970.20.04289-2. Epub 2020 Mar 16. PMID 32181610
- [Result] Miloro M, Criddle TR. Does Low-Level Laser Therapy Affect Recovery of Lingual and Inferior Alveolar Nerve Injuries? J Oral Maxillofac Surg. 2018 Dec;76(12):2669-2675. doi: 10.1016/j.joms.2018.06.001. Epub 2018 Jun 11. PMID 30509397
- [Result] Lomke MA. Clinical applications of dental lasers. Gen Dent. 2009 Jan-Feb;57(1):47-59. PMID 19146143